CLINICAL TRIAL: NCT05434208
Title: Effects of Nurse-led Telephone Based Service for Early Palliative Care Patients With Advanced Cancer: the Paltel Randomized Controlled Trial
Brief Title: Effects of Nurse-led Telephone Based Service for Early Palliative Care (PALTEL)
Acronym: PALTEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRST100.57
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Palliative Care; Cancer
Keywords: Early Palliative Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A RESEARCH ARM: active telephonic follow-up by specialist nurse (Experimental): Early Palliative Care cancer patients will be randomized to active telephonic follow-up program by specialist nurses until end-of-treatment (28 days)
  * Scheduled phone-calls each 7 days from T0 + unscheduled phone-calls (as needed)
    * Questionnaire: ESAS and IPOS;
    * Weight;
    * Medication intake;
    * ECOG-PS
  * Scheduled phone-calls at End of Treatment (28 days from T0):
    * Questionnaire: ESAS and IPOS
    * Questionnaire: FAMCARE-2 for CGs
  Interventions: Other: Nurse-led telephonic calls
- B CONTROL GROUP: face-to-face visit at end of treatment (No Intervention): Early Palliative Care cancer patients will be randomized to face-to-face visit at end of treatment (28 days)
  * Unscheduled phone-calls, on patients initiative:
    * Questionnaire: ESAS and IPOS;
    * Weight;
    * Medication intake;
    * ECOG-PS
  * Face-to-face visit at End of Treatment (28 days from T0):
    * Questionnaire: ESAS and IPOS
    * Questionnaire: FAMCARE-2 for CGs

INTERVENTIONS:
Other: Nurse-led telephonic calls — active telephonic follow-up program by specialist nurses until end-of-treatment (28 days)
  Arms: A RESEARCH ARM: active telephonic follow-up by specialist nurse

SUMMARY:
Non-pharmacological, interventional, two-arm, randomized controlled trial. Early Palliative Care cancer patients will be randomized to active telephonic follow-up program by specialist nurses until end-of-treatment (28 days) (group A, research arm) or face-to-face visit at end of treatment (28 days) (group B, control arm).

There are few studies demonstrating the efficacy of nurse-led telephone service in advanced cancer patients but it's still quite unclear how they can affect quality of life, symptom burden and caregivers distress. In addition, the ideal structure, method and timing of telephone follow-up as well are often not considered and have not been articulated. Nurse-led management by phone to advanced cancer patients could, for some patients, dramatically improve their care experience, quality of life and symptoms control.

Investigators want to build an effective and sustainable approach for implementing the telephone service providing nurse-led telephone-based support to Early Palliative Care cancer patients. The aim is to investigate the feasibility of a proactive approach and measure the efficacy in terms of symptom management, satisfaction with care and impact on health care resources.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study;
* Patients having a defined Caregiver
* Cancer patients referred for the first time to the Early Palliative Care Outpatient Clinic;
* Both Female or Male, aged ≥ 18 years;
* Italian speaking patients.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 3 or higher
* Patients cognitively impaired or deaf;
* Patients not having a telephone or not capable of speaking/using a telephone;
* Patients referred to palliative Homecare or Hospice at the first visit Early Palliative Care Outpatient Clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Edmonton Symptoms Assessments System (ESAS) | 3 years
  ESAS is a questionnaire to rate common symptoms experienced by cancer patients, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being and shortness of breath. The severity at the time of assessment of each symptom is rated from 0 to 10 on a numerical scale, with 0 meaning that the symptom is absent and 10 that it is the worst possible severity (total score 0-90).
Italian Integrated Palliative Care Outcome Scale (IPOS) | 3 years
  The IPOS is a patient-reported outcome measures, valid and reliable both in patient self-report and staff proxy-report versions to assess and monitor symptoms and concerns in advanced illness, determine the impact of healthcare interventions, and demonstrate quality of care.

SECONDARY OUTCOMES:
FAMCARE-2 | 3 years
  The FAMCARE-2 scale includes 17 items and measures caregivers satisfaction with care received by both patent and caregivers with the following four components of care: management of physical symptoms and comfort, provision of information, family support, and patient psychological care. Each item is rated according to a 5-point Likert scale (5=very satisfied - 1=very dissatisfied). The score range is between 17 and 85: high scores indicate high levels of satisfaction with care.
Use of healthcare services | 3 years
  Number of unscheduled hospital admissions, emergency department visits, face-to-face visit in early Palliative Care Outpatient Clinic, unscheduled phone-calls to Palliative Care telephone service for patients or caregivers needs and unscheduled visits in oncological day-hospital. All this data will be collected at End of Study using patients' medical records.
Number of hospital referrals | 3 years
  Number of home care and hospital referrals in group A and B
Patients' access to the local Palliative care network | 3 years
  Mean number of days in home care and hospital in group A and B
Intervention of Palliative Care Outpatient Clinic | 3 years
  Collection of the reasons that led the oncologist to request the intervention of the Palliative Care Outpatient Clinic and categorization of each reson in the subset agreed by international panel on Lancet.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Valenti, Nurse, Study Chair — IRCCS IRST
Locations (1):
- IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l., Meldola, Forlì-Cesena, Italy